CLINICAL TRIAL: NCT04811508
Title: Retrospective Study to Describe Carfilzomib Use on Patients With Relapsed Multiple Myeloma in France in the Context of Carfilzomib Nominative Expanded Access and Compassionate Use
Acronym: CARMYN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Other Study IDs: CHM-2020/S14/07
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2021-03

CONDITIONS: Relapsed Multiple Myeloma
Keywords: relapsed multiple myeloma; Carfilzomib
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective multicenter observational study will provide real-life efficacy and tolerance data for patients with relapsed multiple myeloma (RMM) treated with carfilzomib in the context of nominative expanded access and compassionate use in France, and will allow to evaluate healthcare practices from data obtained during the use of carfilzomib for routine care. Nominative expanded access was open in February 2014 and stopped in march 2016, then relayed by the compassionate program (march 2016- February 2017).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients over the age of 18 years
* Patients beginning carfilzomib treatment in the framework of expanded access or compassionate use in France (KRd or Kd regimen)
* Patients who received carfilzomib in first or second MM relapse
* Patients receiving at least one complete course of carfilzomib

Exclusion Criteria:

* Patients already included in an interventional research protocol using carfilzomib at the time of treatment initiation
* Patients refusing to allow the computerization of their data
* Patients for whom hospital medical records are not accessible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsed multiple myeloma (RMM) treated with carfilzomib in the context of nominative expanded access and compassionate use in France
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Duration of carfilzomib treatment | 31 august 2021
  Assess duration of carfilzomib treatment in adult patients with multiple myeloma who have received carfilzomib at first or second relapse according to the recommendations of the International Myeloma Working Group (time from the date of treatment initiation to the date of permanent discontinuation for any reason)

SECONDARY OUTCOMES:
Time to next treatment | 31 august 2021
  This is defined as the time from the date of treatment initiation (i.e. the date of the first day of the first cycle of the treatment with carfilzomib) to the date when the next line starts. Time to next treatment is censored at the date of death, if applicable. Patients still on carfilzomib treatment at the end of the study will be censored at the date of the last disease evaluation
Progression Free survival (PFS) | 31 august 2021
  Progression free survival is defined as the time from the date of initiation of treatment (i.e. the date of the first day of the first cycle of treatment with carfilzomib) to the date of the first disease progression, as defined by the investigator's judgement using IMWG criteria (1), or the date of death, whichever occurs first. Progression free survival is censored at the date of the last disease evaluation, if applicable

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France